CLINICAL TRIAL: NCT01472055
Title: Pharmacokinetic Study of Fludarabine in Pediatric Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-SCT-1101
Record Dates: First submitted 2011-11-06; First posted 2011-11-16 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Acute Leukemia; Chronic Leukemia; Severe Aplastic Anemia
Keywords: Hematopoietic stem cell transplantation with fludarabine based conditioning
MeSH Terms: conditions — Anemia, Aplastic | interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine (Experimental): Analysis of the pharmacokinetics of fludarabine for hematopoietic stem cell transplantation in pediatric patients
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Fludarabine — 1. Fludarabine 40 mg/m^2 once a day intravenous administration over 30 min
  2. Development of sampling-minimized analysis method through individualized pharmacokinetics Sampling time: 0hr (pre-dose), 30 min (post-dose), 1hr, 3hr, 5hr, 8hr, 24hr
  3. Population pharmacokinetics analysis
  4. Comparative analysis of population pharmacokinetics in pediatric and adult patients
  5. Analysis of population pharmacokinetics, toxicity, engraftment rate, survival rate

SUMMARY:
The purpose of this study is to analysis of the pharmacokinetics of fludarabine for hematopoietic stem cell transplantation in pediatric patients.

DETAILED DESCRIPTION:
Fludarabine is a commonly used chemotherapeutic agent for hematopoietic stem cell transplantation in children. However, no pharmacokinetic study has thus far been conducted in pediatric patients. Fludarabine can cause adverse reactions which include neurotoxicity, damage to lungs. Pharmacokinetic study is critical to predict the safety of fludarabine in pediatric patients.

Through an individualized pharmacokinetic study (which entails numerous samplings) of fludarabine in pediatric patients, this study aims to develop a sampling-minimized analysis method and study the population pharmacokinetics.

Through a pharmacokinetic analysis, we aim to evaluate whether pediatric patients show similar population pharmacokinetics of adults, for whom fludarabine is authorized, and evaluate the safety (toxicity) and efficacy (event free survival).

ELIGIBILITY:
Inclusion Criteria:

1. Conditioning regimen including fludarabine
2. Age: < 19 years old
3. Functional class: ECOG 0-2
4. No loss of function of major organs. Criteria may be individualized.

   * Heart: shortening fraction > 30%, ejection fraction > 45%.
   * Liver: total bilirubin < 2 ⅹ upper limit of normal; ALT < 3 ⅹ upper limit of normal.
   * Kidney: creatinine < 2 ⅹ normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
5. No active viral or fungal infection
6. Appropriate hematopoietic stem cell donor
7. Informed consent from patients' parents

Exclusion Criteria:

1. Pregnant or breast feeding
2. Disease progression due to clinical test
3. Psychiatric disease may interfere with clinical test
4. Whether attending physician consider the patient inappropriate for study enrollment

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of the pharmacokinetics of fludarabine for hematopoietic stem cell transplantation in pediatric patients | 0hr (pre-dose), 30 min, 1, 3, 5, 8, 24hrs post-dose

SECONDARY OUTCOMES:
Comparative analysis of the pharmacokinetics of fludarabine in pediatric and adult patients | 3 years
Evaluation of toxicity, event free survival according to the pharmacokinetics of fludarabine | 1, 3, 6 and 12 months after transplantation
Evaluation of therapy related toxicity, significant adverse reaction | for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehangno, Jongno-gu, South Korea